CLINICAL TRIAL: NCT04499872
Title: Planning for Future Care With Patients With Advanced Cancer: Examining the Feasibility of Using the Trajectory Touchpoint Technique for Advance Care Planning.
Brief Title: Planning for Future Care With Patients With Advanced Cancer
Status: Completed | Type: Observational
Sponsor: Liverpool University Hospitals NHS Foundation Trust (Other Government)
Collaborators: University of Liverpool (Other)
Responsible Party: Sponsor
Other Study IDs: RLBUHT5869; 261984 (Other: HRA)
Record Dates: First submitted 2019-06-21; First posted 2020-08-05 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2019-06

CONDITIONS: Advance Care Planning
Keywords: Palliative care

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient/family Participant: Advance Care Plan with the Trajectory Touchpoint Technique
  Interventions: Other: Advance Care Plan with Trajectory Touchpoint Technique

INTERVENTIONS:
Other: Advance Care Plan with Trajectory Touchpoint Technique — Advance Care Plan with Trajectory Touchpoint Technique
  Other Names: ACP TTT

SUMMARY:
Advance Care Planning (ACP) is a process where patients (and their families if appropriate) discuss with their doctors and nurses what may happen as their illness progresses, including how they (and their family) would like to be supported and cared for. The discussion of expectations and choices for care can then be formally recorded and used to guide and inform future care. Well documented benefits of ACP include empowering patients and their families to better understand available choices and make informed decisions regarding future care; This ensures care is based on what is important to that patient (and their family) and prepares all for the end of life. However, few people with a life limiting illness (such as cancer) have an ACP. Patients and families often find future and end of life care a difficult subject to discuss, as do doctors/nurses, who fear upsetting patients and families and who may have limited training/experience in how to prompt and record ACP discussions.

This project aims to overcome the barriers in discussing ACP by using the Trajectory Touchpoint Technique. The technique utilises a range of existing service evaluation and service design methods found in "service management" and "design systems". Rich pictures are used in the form of cartoons on an electronic tablet or printed card, to enable patients/families to lead discussions. The images are simple and enable people to raise sensitive and potentially distressing topics at a pace they are comfortable with, rather than responding to numerous pre-determined questions. The technique was originally designed to explore the experiences of patients (and their families) of Hospice Care and has been successfully used in over 200 interviews, demonstrating an ability to sensitively facilitate difficult conversations whilst enabling rich and detailed discussion.

DETAILED DESCRIPTION:
1.1 BACKGROUND In 2014, academics at the University of Liverpool Management School who are service quality researchers were approached by East Cheshire Hospice (ECH). ECH provides specialist palliative care for people with progressive life-limiting illnesses, providing services to patients, carers and families via inpatient and outpatient units and day facilities. ECH strives for excellence in service and the patient experience. Anecdotal stories and other forms of feedback provided plenty of evidence that the work of the hospice was meaningful. However, ECH did not have any systematic, robust way of capturing these experiences. Hence, while ECH was often told it had transformed the experience of patient's at the most critical time in their lives and that it was needed and appreciated by many service users, there was nothing but anecdotal evidence to back up this feedback. Worried that such superb feedback could actually lead to complacency, the team at ECH commissioned the University to undertake a 'deep-dive' of the impact of hospice services upon the different inpatient and outpatient service users associated with ECH.

The team, comprising Prof Philippa Hunter-Jones and Dr. Lynn Sudbury-Riley, designed a new qualitative research technique to follow the user's experience at every touchpoint in their journey. In 2015, interviews with 38 in-patients, outpatients, visitors and bereaved families enabled a 'deep-dive' to uncover perceptions of the whole service experience among these diverse users. Results of this new approach suggested the technique fully captures the hospice experience and suggests areas for improvements to hospice services. Indeed, the results of the study have informed the strategy and operations of ECH, and, mindful of continuous improvement, ECH have requested that the exercise is repeated.

Other hospices heard of the success of this work and the team were commissioned by Oakhaven Hospice in Hampshire to work with them, too. Additionally, based on the success of the project, the project was shortlisted by the school for a REF impact case, and the team were awarded funding to repeat the project in further hospice and palliative care settings.

The Academic Palliative Care Unit on 4Y at RLBUHT was one of the palliative care units to be evaluated next. From the service evaluation project on 4Y grew the novel idea to use the TTT as part of the Advanced Care Planning (ACP) conversation lead by clinicians. ACP is not consistently carried out for all patients that might have a need. There is also not a consistent way in which ACP is conducted to ensure quality is maintained within the patient centric approach.

1.2 RATIONALE FOR CURRENT STUDY Advance Care Planning (ACP) is the process of making choices and plans in regards of future care for patients with life limiting disease, particularly those who may lose the capacity to communicate. ACP has been shown to positively impact on the quality of end-of-life care, yet few (only 6-8%) have a completed formal ACP: a result of patients' anxieties about discussing future care issues and clinicians' concerns over responsibility and starting a "difficult" conversation.

This project will test a new methodology, the Trajectory Touchpoint Technique - a visual/pictorial technique - that aids difficult conversation. In a recent trial, the technique has successfully enabled patients to direct in-depth and sensitive conversations regarding their experiences of Hospice care. This technique exhibits the potential to overcome barriers in ACP discussions, enabling patients to direct the conversation at their pace/level of comfort, and empowering clinicians to sensitively facilitate depth and detail. Therefore the research question is: Is the Trajectory Touchpoint Technique a feasible intervention to support Advance Care Planning in patients/families with advanced cancer.

1.3 THE TRAJECTORY TOUCHPOINT TECHNIQUE The Trajectory Touchpoint Technique uses the concept of touchpoints; anything that fosters or impacts experiences. Touchpoints are any potentially important issue that a participant may wish to talk about. It is important to stress that a touchpoint is only valid if it is considered to be so by the participant. Potential touchpoints can be big or small, tangible or intangible. Rich pictures, in the form of cartoons and easy to recognise signs and symbols are used to reference potentially important touchpoints. Such rich picture methodologies are particularly appropriate for complex research situations where multiple forces and interactions between those forces are present, and can capture and elucidate potential influences that may otherwise remain hidden.

The technique uses a qualitative, narrative data collection method and touchpoints are grouped together into key stages or themes. These groups of cartoon touchpoints are presented on an I-Pad/Electronic Tablet or printed onto large laminated cards and used as a prompt/aide memoire to guide discussion. Figure 1 provides an example of one group of touchpoints used to collect data on the experiences of care in a children's hospice.

Prior use of the technique with over 200 palliative care patients and their families demonstrates that the cartoons make people smile and help people to relax, even when the content of the discussion is distressing. Patients and their families are free to choose from the range of touchpoints, and to add anything else that they may see fit. Importantly, the pictures guide the discussion, making difficult discussions easier as there is a greatly reduced need for probing and/or pre-determined clinician led questioning. Touchpoints remind people of things that they may have otherwise omitted from the discussion. Our experience suggests that the technique enables a 'deep dive' into the feelings, fears and wishes of palliative care patients and their families, aids systematic and comprehensive data collection, yet is very easy to use and understand.

ELIGIBILITY:
Inclusion Criteria:

* Cared for on the Academic Palliative Care Unit
* Diagnosis of Cancer
* No Advance Care Plan (or ACP needs updating)
* Able to provide informed consent (has capacity)

Exclusion Criteria:

* Absence of cancer
* Has current ACP
* Deemed to unwell by the APCU MDT
* Unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who could benefit from an ACP discussion and are located on ward 4Y of the Academic Palliative Care Unit of Royal Liverpool Broardgreen University Hospital NHS Trust.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2019-07-10 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Interview question: please share in your own words your opinion of the ACP discussion | within 72 hours of consent.
  Participant is asked to join a 1:1 interview discussion. VERBAL DIALOGUE NO SCALE they talk about their ACP. Thematic Analysis will be conducted on the interview transcript to understand the common themes raised throughout the different interviews.

CONTACTS AND LOCATIONS:
Overall Officials: Professor, Study Chair — Royal Liverpool Broadgreen University Hospital NHS Trust
Locations (1):
- Liverpool University Hospitals NHS Foundation Trust, Liverpool, Merseyside, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
data will be anonymised and archived for use in other research projects in the future. After 10 years all data will be destroyed.
Supporting Information: CSR
Time Frame: Within 3 months of study completion
Access Criteria: Only the named investigators will have access to the data.

DOCUMENTS (1):
  • Study Protocol (2020-02-01): https://cdn.clinicaltrials.gov/large-docs/72/NCT04499872/Prot_000.pdf